CLINICAL TRIAL: NCT06989970
Title: Treating Traumatic Brain Injury With Transcranial Direct Current Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Ybrain Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00353047
Record Dates: First submitted 2025-04-30; First posted 2025-05-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Traumatic Brain Injury; Chronic Traumatic Brain Injury; transcranial direct current stimulation; tDCS; Computerized Cognitive Therapy
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: This is a repeated measures crossover trial, where all participants will receive dorsolateral prefrontal cortex (DLCPFC) stimulation followed by sham stimulation or vice versa. Each condition will be separated by 2 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both interventions, whether involving tDCS or sham stimulation, will entail a gradual increase in electrical current at the commencement of the stimulation, inducing a transient tingling sensation on the scalp that typically dissipates within seconds. While the ramping process necessitates input from the researcher, it is now feasible to implement blinding procedures for study staff administering tDCS and participants. This is facilitated by a device that enables another team member to designate the setting as "tDCS" or "sham" without the therapist's knowledge. Following the ramping phase, in the sham condition, the intensity of stimulation decreases to 0 mA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS on the DLPFC + Cognitive Intervention(s) then Sham tDCS (Active Comparator): Participants will receive left DLPFC active tDCS for 3 weeks, followed by a follow-up immediately after and 2 months later. Active tDCS will be administered for 20 minutes. Cognitive training exercises will be administered concurrently with the tDCS and will take approximately 40 minutes to complete.
  Interventions: Combination Product: Active tDCS on the DLPFC + Cognitive Intervention(s); Combination Product: Sham tDCS on the DLPFC + Cognitive Intervention(s)
- Sham tDCS on the DLPFC + Cognitive Intervention(s) then Active tDCS (Sham Comparator): Participants will receive left DLPFC active tDCS for 3 weeks, followed by a follow-up immediately after and 2 months later. Cognitive training exercises will be administered concurrently with the sham tDCS and will take approximately 40 minutes to complete
  Interventions: Combination Product: Active tDCS on the DLPFC + Cognitive Intervention(s); Combination Product: Sham tDCS on the DLPFC + Cognitive Intervention(s)

INTERVENTIONS:
Combination Product: Active tDCS on the DLPFC + Cognitive Intervention(s) — Combination Product: Active tDCS and cognitive training intervention. Participants will receive cognitive training paired with active tDCS for 3 weeks, followed by follow-up sessions immediately after and 2 months later, during which the patient's performance on the cognitive training exercises and executive functions will be assessed. Cognitive training exercises have been drawn from a computer-aided cognitive training program (BrainHQ).
  For the active tDCS, stimulation will be delivered by a battery-driven constant current stimulator. The electrical current will be administered to the left DLPFC at an intensity of 2 milliamperes (mA) (estimated current density 0.04 mA/cm2; estimated total charge 0.048 Coulombs/cm2) in a ramp-like fashion for a maximum of 20 minutes.
Combination Product: Sham tDCS on the DLPFC + Cognitive Intervention(s) — Combination Product: Sham tDCS and cognitive training intervention
  Participants will receive cognitive training paired with sham tDCS for 3 weeks, followed follow-up sessions immediately after and 2 months later, during which the patient's performance on the cognitive training exercises and executive functions will be assessed. Cognitive training exercises have been drawn from a computer-aided cognitive training program (BrainHQ).
  For the sham tDCS, electrodes will be placed in the same area as in the active tDCS condition, but current will be administered in a ramp-like fashion but after the ramping the intensity will drop to 0 mA. Current under the Sham condition will last for a maximum of 30 seconds.

SUMMARY:
Traumatic Brain Injury (TBI) often results in a wide array of cognitive impairments, which can significantly diminish quality of life for affected individuals. While traditional rehabilitation methods typically adopt a standardized approach, it's crucial to acknowledge the significant heterogeneity within the TBI patient population. Neglecting these variations reduces the likelihood of otherwise effective treatments being considered for widespread adoption. Emerging evidence highlights the potential of transcranial direct current stimulation (tDCS) as a promising adjunctive therapy. tDCS, a noninvasive and safe neuro-rehabilitative procedure, has shown efficacy when integrated with cognitive training across various neurological disorders, such as depression, post-stroke aphasia, and neurodegenerative conditions.

This study aims to investigate the effectiveness of tDCS paired with behavioral therapy, particularly cognitive training, in improving cognition and executive function in chronic TBI patients. Additionally, tDCs targets in the current study will be tailored to each individual patient, recognizing the patient's unique needs and circumstances

DETAILED DESCRIPTION:
Objective: This pilot study (targeting a sample of 10 TBI patients) aims to investigate whether combining cognitive training with anodal tDCS can enhance cognitive function more effectively compared to cognitive training alone in individuals with chronic TBI. The target for tDCS application will be the left dorsolateral prefrontal cortex (DLPFC), thought to be the area associated with executive impairment in TBI patients.

Study Design: Each participant will undergo an initial neuropsychological evaluation and Functional magnetic resonance imaging (fMRI). Following the preliminary evaluation, participants will undergo either tDCS or sham stimulation for 3 weeks, with follow-up assessments immediately after and 2 months later, to measure cognitive training progress. After the 2-month follow-up, participants will undergo another 3 weeks of cognitive training with either sham or tDCS, based on the participant's condition in phase 1. Post-training, there will be additional follow-ups immediately after and 2 months later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of traumatic brain injury (TBI) at least 2 years prior to participation
* Right-handed
* English - speaking

Exclusion Criteria:

* Uncorrected visual impairment
* Uncorrected hearing impairment
* Stroke or other premorbid neurological disorders affecting the brain
* Premorbid learning disorders

MRI Exclusion Criteria:

* severe claustrophobia
* Cardiac pacemakers, ferromagnetic implants, cochlear implants
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2029-10-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in Selective attention and cognitive flexibility as assessed by the Attention Network Task (ANT) | Before intervention, immediately after intervention
  This will be measured using the Attention Network Task (ANT). An efficiency score for executive attention is derived by comparing scores on trials with congruent flankers to trials with incongruent flankers. Subjects will tend to be slower and less accurate for incongruent trials, the size of the difference indicates the extent to which an individual can supress conflicting response tendencies. A larger difference between congruent and incongruent trials score indicates a lower executive efficiency (score range: 0-96)..
Change in attention and task switching as assessed by the N-Back score | Before intervention, immediately after intervention
  The N-back task is a well-established task that assesses working memory and working memory capacity. Participants are presented with words in sequence and instructed to reply whether the current word matches the one presented 2 words ago (2-back). Scoring will be based on the total number of correct responses (hit rate) minus the number of incorrect responses (false alarm rate), where a greater score is better (score range: 0-80).
Change in Self-Ordered Pointing Task (SOPT) | Before intervention, immediately after intervention
  The SOPT is a test used to assess executive functioning. In this task, participants are shown a series of pages, each displaying the same set of abstract images arranged in a random order. On each page, the participant must point to one image, ensuring not to select the same image more than once across the entire series. A correct response involves selecting a previously un-chosen image, while an error is recorded when a participant selects an image already chosen on a previous page. Performance will be measured by total number of errors measured out of the total number of possible responses, with a higher error count indicating greater impairment.

SECONDARY OUTCOMES:
Change in attention and task switching as assessed by the Trail Making Task | Before intervention, immediately after intervention
  This will be measured using Trail Making Task and N-Back scores. The Trail Making Test is scored by time. Participants are allowed 0 - 300 seconds to complete the task. Less time needed to complete the task is indicative of better task-switching.
Change in Digit Span Forward | Before intervention, immediately after intervention
  Digit span forward involves the recall of a series of single digits (sets of 1-8 digits) in the same order the digits were presented. Scoring is based on the number of digits or blocks shown in a trial (i.e. 1,7 is 2 digits). There are two trials for each span, if both trials are correct the score is a whole number (i.e. 2). If one trial is incorrect in a span, subtract 0.5 from that tier (i.e. 1.5). A higher number is considered better. (Score range for forward tasks: 0-9)
Change in Digit Span Backward | Before intervention, immediately after intervention
  This will be measured using Digit Span Backward for verbal working memory and spatial span Backward for spatial working memory. The digit span backward is a well-established task that assesses rote immediate verbal memory and working memory. Participants are presented with a series of digits and are instructed to repeat the digits in the reverse order. Scoring is based on the number of digits shown in a trial (i.e. 1,7 is 2 digits). There are two trials for each span, if both trials are correct the score is a whole number (i.e. 2). If one trial is incorrect in a span, subtract 0.5 from that tier (i.e. 1.5). A higher number is considered better. (Score range for backwards tasks: 0-8)
Change in attention and inhibition as assessed by the Simon Task | Before intervention, immediately after intervention
  This will be measured using Simon test scores. The Simon task assesses an individual's ability to flexibly shift the perceptual focus in response to changing demands, particularly the participant's capacity to inhibit a habitual response in favor of an unconventional one. Performance on the Simon task is typically scored based on measures such as reaction time and accuracy. Increased reaction times and higher error rates on incongruent trials are indicative of greater difficulty in inhibiting the interference caused by the word's meaning, reflecting decreased cognitive flexibility and inhibition abilities (accuracy score range: 0-120).
Change in Spatial Span Forward | Before intervention, immediately after intervention
  Spatial span forward involves the recall of a series of of positions on a board (sets of 1-9) in the same order the digits were presented. Scoring is based on the number of blocks shown in a trial (i.e. 1,7 is 2 blocks). There are two trials for each span, if both trials are correct the score is a whole number (i.e. 2). If one trial is incorrect in a span, subtract 0.5 from that tier (i.e. 1.5). A higher number is considered better. (Score range for forward tasks: 0-9)
Change in Spatial Span Backward | Before intervention, immediately after intervention
  This will be measured using Spatial Span Backward. Participants are presented with a series of block positions and are instructed to repeat the positions in the reverse order. Scoring is based on the number of blocks shown in a trial (i.e. 1,7 is 2 blocks). There are two trials for each span, if both trials are correct the score is a whole number (i.e. 2). If one trial is incorrect in a span, subtract 0.5 from that tier (i.e. 1.5). A higher number is considered better. (Score range for backwards tasks: 0-8)

OTHER OUTCOMES:
Change in Global Cognitive Scores as assessed by the Montreal Cognitive Assessment (MoCA) | Before intervention, immediately after intervention
  This will be measured using the Montreal Cognitive Assessment (MoCA). Scored from 0-30 points, higher is better.
Change in verbal fluency task score | Before intervention, immediately after intervention
  Verbal fluency tasks (semantic and letter fluency) involve generating as many words as possible in one minute. Scoring will be based on number of words generated per minute. The investigators will compute the raw score of items correct and compute change in outcome between baseline and each time point. Increase in score is considered benefit.
Change in semantic content of connected speech | Before intervention, immediately after intervention
  Using the Cookie Theft image from the Boston Diagnostic Aphasia Examination (BDAE) investigators will obtain representative language samples as participants describe the images. The investigators will compute the raw score of items (semantics) correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in spelling as assessed by the Johns Hopkins Dysgraphia battery | Before intervention, immediately after intervention
  Accuracy in spelling using the Johns Hopkins Dysgraphia battery will be compared for tDCS and sham conditions. The investigators will compute the raw score of items correct using a spelling scoring system accounting for additions, substitutions, and deletions. Each word will get a score from 0-1 and the average of pseudowords and real words will be computed and transformed to percent correct (range: 0-100%), computing change in outcome in percent difference before intervention and each time point after. Increase in score is considered a benefit.
Change in Oral Naming as assessed by Boston Naming Test score | Before intervention, immediately after intervention
  Accuracy in oral picture naming (30-item Boston Naming Test) will be compared for tDCS and sham conditions. The Boston Naming Test is a widely used picture naming test that detects lexical retrieval deficits in the oral modality. The investigators will compute the raw score of items correct (range 0-30 items) and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Kyrana Tsapkini, PhD., Principal Investigator — Johns Hopkins University